CLINICAL TRIAL: NCT01710813
Title: A Prospective Safety Sub-Registry to Assess Anaphylaxis and Severe Allergic Reactions, and Severe Cutaneous and Systemic Immune Complex Mediated Reactions With Alglucosidase Alfa Treatment
Brief Title: Alglucosidase Alfa Pompe Safety Sub-Registry
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AGLU06909; LTS13930 (Other: Other company study code)
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Pompe Disease
Keywords: pompe disease; alglucosidase alfa; anaphylaxis; severe cutaneous; systemic immune complex-mediated reactions
MeSH Terms: conditions — Glycogen Storage Disease Type II; Anaphylaxis | interventions — GAA protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pompe safety sub-registry: patients are selected from those who are enrolled in the Pompe Registry, and will be followed for safety evaluation in this sub-registry
  Interventions: Biological: alglucosidase alfa

INTERVENTIONS:
Biological: alglucosidase alfa — Alglucosidase alfa IV infusion of 20 mg/kg; qow
  Other Names: Myozyme; Lumizyme

SUMMARY:
To collect uniform and meaningful data on patients with Pompe disease who experience anaphylaxis, severe allergic reactions, and/or signals of severe cutaneous and/or systemic immune complex-mediated reactions following treatment with alglucosidase alfa.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be enrolled in the Pompe Registry;
* Provide a signed patient information and authorization form;
* Have a confirmed diagnosis of Pompe disease (confirmation of diagnosis is defined as documented GAA enzyme deficiency from any tissue source and/or documentation of 2 GAA gene mutations);
* Be naïve to and plan to be treated with alglucosidase alfa at or prior to enrollment, or are being treated with alglucosidase alfa.

Exclusion Criteria:

* Patients will be excluded if they have received an investigational drug (excluding alglucosidase alfa) within 30 days prior to signing a Safety Sub-Registry Patient Information and Authorization form, or if they are taking or plan to take any investigational product while enrolled in the Safety Sub-Registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are enrolled in the Pompe Registry will be enrolled in this sub-registry include patients with infantile-onset Pompe disease, as well as those with late-onset Pompe disease.
  An approximately equal proportion of currently treated and treatment-naïve patients is targeted for enrollment at each site.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
number of patients experience anaphylaxis, severe allergic reactions and/or signals of severe cutaneous and/or systematic immune complex-mediated reactions | 4 Years
  collect meaningful data on patients with these outcomes following treatment with alglucosidase alfa

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (18):
- United States (6):
  - Investigational Site Number 840016, Phoenix, Arizona
  - Investigational Site Number 840002, Durham, North Carolina
  - Investigational Site Number 840004, Hershey, Pennsylvania
  - Investigational Site Number 840014, Pittsburgh, Pennsylvania
  - Investigational Site Number 840008, Salt Lake City, Utah
  - Investigational Site Number 840001, Fairfax, Virginia
- Belgium (3):
  - Investigational Site Number 056001, Ghent
  - Investigational Site Number 056002, Leuven
  - Investigational Site Number 056003, Leuven
- Investigational Site Number 203001, Prague, Czechia
- Investigational Site Number 276002, Halle, Germany
- Italy (6):
  - Investigational Site Number 380001, Brescia
  - Investigational Site Number 380002, Cagliari
  - Investigational Site Number 380006, Messina
  - Investigational Site Number 380005, Milan
  - Investigational Site Number 380004, Padua
  - Investigational Site Number 380003, Roma
- Investigational Site Number 158001, Taipei, Taiwan